CLINICAL TRIAL: NCT05943327
Title: Interventional, Randomized, Double-blind, Sequential Cohort, Placebo-controlled, Multiple-dose Trial Investigating the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Properties of Lu AG06474 in Healthy Young Men and Women, With an Open-label, Cross-over, Single-dose Part Investigating the Relative Bioavailability of a Capsule Formulation
Brief Title: A Study Investigating Lu AG06474 in Healthy Young Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: For strategic reasons
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20065A
Record Dates: First submitted 2023-06-16; First posted 2023-07-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Multiple Doses of Lu AG06474 or Placebo (Experimental): Participants will receive multiple oral doses of Lu AG06474 or placebo.
  Interventions: Drug: Lu AG06474; Drug: Placebo
- Part B: Single Doses of Lu AG06474 (Experimental): Participants will receive single oral doses of Lu AG06474.
  Interventions: Drug: Lu AG06474

INTERVENTIONS:
Drug: Lu AG06474 — Oral Solution
Drug: Placebo — Oral Solution
  Arms: Part A: Multiple Doses of Lu AG06474 or Placebo
Drug: Lu AG06474 — Capsule
  Arms: Part B: Single Doses of Lu AG06474

SUMMARY:
The purpose of this study is to investigate the safety of multiple oral doses of Lu AG06474, how well the doses are tolerated, and what the body does to the drug after administering it to healthy young participants. This study also aims to compare how the body absorbs and uses Lu AG06474 when it is given in capsule form versus when it is given as an oral solution.

DETAILED DESCRIPTION:
The study has 2 parts: Part A and Part B.

Part A consists of up to 7 sequential cohorts (Cohorts A1 to A7), with 8 participants per cohort randomized to receive multiple doses of either Lu AG06474 or placebo: 6 will receive Lu AG06474 oral solution and 2 will receive placebo.

Part B consists of 1 cohort (Cohort B1), with 12 participants: all participants will receive 2 single doses of Lu AG06474 (one as an oral solution and one in capsule form), taken 3 days apart.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30 kilograms per meter squared (kg/m^2) at the Screening Visit and at the Baseline Visit.
* The participant has a resting supine pulse ≥50 and ≤100 beats per minute (bpm) at the Screening Visit and at the Baseline Visit. For physically/athletically well-trained participants, the lower limit is ≥45 bpm.
* The participant has a resting supine systolic blood pressure ≥91 and ≤140 millimeters of mercury (mmHg) and a resting supine diastolic blood pressure ≥51 and ≤85 mmHg at the Screening Visit and at the Baseline Visit.

Exclusion Criteria:

* The participant has previously been dosed with Lu AG06474.
* The participant has participated in a clinical trial <30 days prior to the Screening Visit.
* The participant has taken any investigational medicinal product ≥30 days or <5 half-lives of that product, whichever is longer, prior to the first dose of IMP.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants with Treatment Emergent Adverse Events (AEs) | Up to Day 10
Part A: Electrocardiogram (ECG) Parameter (delta QTcF) on Day 5 | Day 5
Part A: AUC0-τ: Area Under the Lu AG06474 Plasma Concentration Curve During Dosing Interval | Predose to Day 7
Parts A and B: Cmax: Maximum Observed Plasma Concentration of Lu AG06474 | Predose to Day 6
Parts A and B: Tmax: Nominal Time Corresponding to the Occurrence of Cmax | Predose to Day 6
Parts A and B: t½: Apparent Elimination Half-life of Lu AG06474 | Predose to Day 6
Part B: AUC0-infinity: Area Under the Lu AG06474 Plasma Concentration Curve From Zero to Infinity | Predose to Day 6
Part A: Accumulation Index | Predose to Day 7
Part B: Frel: Relative Bioavailability | Predose to Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Miami, Miami, Florida, United States